CLINICAL TRIAL: NCT06640296
Title: Tolerability and Effectiveness of Extended Dosing of Liposomal Amphotericin B (L-AmB) for Primary Prophylaxis of Invasive Fungal Disease in High-risk Pediatric Patients: a Retrospective Multicenter Study
Brief Title: L-AmB_ Retrospective mUlticenter Study on Mycosis prOphylaxis
Acronym: L-AmB_RUSCO
Status: Enrolling by invitation | Type: Observational
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Elio Castagnola, MD, Istituto Giannina Gaslini
Other Study IDs: N. CET Liguria 366/2023
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Invasive Fungal Infections; Prophylaxis; Invasive Fungal Disease
MeSH Terms: conditions — Invasive Fungal Infections | interventions — liposomal amphotericin B

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Patients at high risk of developing IFD: patients at high risk of developing IFD receiving chemotherapy for (1st line or relapse treatment) or allo-HSCT for which primary fungal prophylaxis with Liposomal amphotericin B has been administered between 01/01/2019 to 31/12/2023
  Interventions: Drug: Liposomal Amphotericin B (LAmB)

INTERVENTIONS:
Drug: Liposomal Amphotericin B (LAmB) — collect data on tolerability and effectiveness of liposomal amphotericin B prophylaxis

SUMMARY:
Invasive fungal disease (IFD) still represents an important cause of morbidity and mortality in immunocompromised patients, particularly in patients undergoing antineoplastic chemotherapy or allogeneic hemopoietic stem cell transplantation (allo-HSCT). International guidelines recommend primary antifungal prophylaxis to reduce mortality and morbidity in these patients. Liposomal amphotericin B (L-AmB) can represent a valid alternative for antifungal prophylaxis in pediatric age as its spectrum is extended to both molds and yeasts, has reduced pharmacological interactions with the antineoplastic drugs most frequently used in treatment protocols. All this despite the availability of an intravenous formulation which can ensure complete compliance with the treatment. L-AmB prophylaxis has been proposed with different dosages: 1 mg/kg every other day vs 2.5 mg/kg/dose twice-a-week vs 5 mg/kg/once-a-week)

DETAILED DESCRIPTION:
Invasive fungal disease (IFD) still represents an important cause of morbidity and mortality in immunocompromised patients, particularly in patients undergoing antineoplastic chemotherapy or allogeneic hemopoietic stem cell transplantation (allo-HSCT). In this setting children presents some differences compared to adults in terms of risk factors for IFD: different treatment schemes, age-related comorbidities, diagnostic tools with different sensitivity. International guidelines strongly recommend primary prophylaxis in children at high risk of developing IFD to reduce disease-related morbidity and mortality (patients are considered to be at high risk in the presence of an IFD incidence ≥10%). Although the risk factors are well characterized in the literature and substantially unchanged over time, the local epidemiology must be considered in the evaluation of the best prophylaxis strategy. Drugs presently recommended for antifungal prophylaxis have been poorly studied in children, anyway triazoles (mainly posaconaozle) are indicated as possible prophylactic agents also in pediatrics. However, these drugs can present important interactions with drugs important for the treatment of pediatric leukemias (e.g. vinca alkaloids and posaconazole) and sometimes they lack of specific pediatric formulations, fact that can reduce compliance because of bad taste of the available formulations (oral solutions) or difficulties in swallowing and risk of poor absorption in presence of mucositis (bulky, non-divisible pills or capsules). Liposomal amphotericin B (L-AmB) can represent a valid alternative for antifungal prophylaxis in pediatric age as its spectrum is extended to both molds and yeasts, has reduced pharmacological interactions with the antineoplastic drugs most frequently used in treatment protocols. All this despite the availability of an intravenous formulation only which may require hospital access or activation of the home care team, but which can ensure complete compliance with the treatment. L-AmB prophylaxis has been proposed with different dosages: 1 mg/kg every other day vs 2.5 mg/kg/dose twice-a-week vs 5 mg/kg/once-a-week).

ELIGIBILITY:
Inclusion Criteria:

* all patients at high risk of developing IFD receiving chemotherapy for (1st line or relapse treatment) or allo-HSCT for which primary fungal prophylaxis with extended dosing of liposomal amphotericin B has been administered

Exclusion Criteria:

* previous diagnosis of IFD (secondary prophylaxis),
* contraindications to liposomal amphotericin B prophylaxis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients who received extended dosing of liposomal amphotericin B prophylaxis from 01/01/2019 to 31/12/2023
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability of extended dosing of liposomal amphotericin B | In the period between the first and last administration of L-AmB
  Number of participants with treatment-related adverse events (both clinical and laboratoristic adverse events) as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Effectiveness of extended dosing of liposomal amphotericin B | Up to 6 months after the last administration of L-AmB
  Number of new diagnoses of IFD classified as proven, probable or possible according to EORTC/MSG criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Giannina Gaslini, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Donnelly JP, Chen SC, Kauffman CA, Steinbach WJ, Baddley JW, Verweij PE, Clancy CJ, Wingard JR, Lockhart SR, Groll AH, Sorrell TC, Bassetti M, Akan H, Alexander BD, Andes D, Azoulay E, Bialek R, Bradsher RW, Bretagne S, Calandra T, Caliendo AM, Castagnola E, Cruciani M, Cuenca-Estrella M, Decker CF, Desai SR, Fisher B, Harrison T, Heussel CP, Jensen HE, Kibbler CC, Kontoyiannis DP, Kullberg BJ, Lagrou K, Lamoth F, Lehrnbecher T, Loeffler J, Lortholary O, Maertens J, Marchetti O, Marr KA, Masur H, Meis JF, Morrisey CO, Nucci M, Ostrosky-Zeichner L, Pagano L, Patterson TF, Perfect JR, Racil Z, Roilides E, Ruhnke M, Prokop CS, Shoham S, Slavin MA, Stevens DA, Thompson GR, Vazquez JA, Viscoli C, Walsh TJ, Warris A, Wheat LJ, White PL, Zaoutis TE, Pappas PG. Revision and Update of the Consensus Definitions of Invasive Fungal Disease From the European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium. Clin Infect Dis. 2020 Sep 12;71(6):1367-1376. doi: 10.1093/cid/ciz1008. PMID 31802125
- [Background] Bochennek K, Tramsen L, Schedler N, Becker M, Klingebiel T, Groll AH, Lehrnbecher T. Liposomal amphotericin B twice weekly as antifungal prophylaxis in paediatric haematological malignancy patients. Clin Microbiol Infect. 2011 Dec;17(12):1868-74. doi: 10.1111/j.1469-0691.2011.03483.x. Epub 2011 Sep 6. PMID 21895857
- [Background] Groll AH, Pana D, Lanternier F, Mesini A, Ammann RA, Averbuch D, Castagnola E, Cesaro S, Engelhard D, Garcia-Vidal C, Kanerva J, Ritz N, Roilides E, Styczynski J, Warris A, Lehrnbecher T; 8th European Conference on Infections in Leukaemia. 8th European Conference on Infections in Leukaemia: 2020 guidelines for the diagnosis, prevention, and treatment of invasive fungal diseases in paediatric patients with cancer or post-haematopoietic cell transplantation. Lancet Oncol. 2021 Jun;22(6):e254-e269. doi: 10.1016/S1470-2045(20)30723-3. Epub 2021 Mar 31. PMID 33811813
- See also: dictionary of the "Common Terminology Criteria for Adverse Events" of the National Cancer Institute — https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_6